CLINICAL TRIAL: NCT06950684
Title: The Effect of Protein Supplementation and Resistance Training on Body Composition, Functional Parameters, Metabolic Adaptation, and Nitrogen Balance in Adults (Aged ≥45 Years) With Overweight/Obesity Receiving Incretin-Based Weight Loss Medication for 6 Months: A Multicenter RCT
Brief Title: Impact of Protein Supplementation and Resistance Training on Body Composition, Functional Parameters, Metabolic Adaptation, and Nitrogen Balance in Adults Aged 45 Years and Older With Overweight or Obesity Receiving Incretin-based Medications
Acronym: PRIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Ariel University (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Dietitian and Epidemiologist, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASMC 0035-25 and TLV-0168-25; 1001829006 (Other Grant/Funding Number: Israel Ministry of Innovation, Science & Technology)
Record Dates: First submitted 2025-04-08; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Overweight (BMI > 25); Weight Loss
Keywords: Protein supplementation; Resistance training; Body composition; Metabolic rate; Nitrogen balance; Incretin-based medications; Wegovy; Mounjaro; Older adults; Obesity treatment
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein Supplementation and Resistance Training (Experimental): Participants in this arm will consume a daily dietary supplement of 25 grams of whey protein powder (Easy Whey) and participate in a structured resistance training program consisting of one guided online session per week, plus two additional independent sessions weekly, for a total duration of 6 months.
  Interventions: Dietary Supplement: Whey Protein Supplement; Behavioral: Resistance Training Program
- Control Group (No Intervention): Participants in this arm will not receive protein supplementation or structured resistance training. They will be provided with general dietary recommendations at the beginning of the study and will continue their usual care for 6 months

INTERVENTIONS:
Dietary Supplement: Whey Protein Supplement — Participants will take a daily supplement of whey protein powder (Easy Whey) providing 25 grams of protein each day for the duration of 6 months
  Arms: Protein Supplementation and Resistance Training
Behavioral: Resistance Training Program — Participants will engage in resistance training consisting of one guided online session each week and two additional independent resistance training sessions weekly, totaling three sessions per week, for a duration of 6 months.
  Arms: Protein Supplementation and Resistance Training

SUMMARY:
This study aim to evaluate the effects of protein supplements and resistance training on body composition, functional parameters, metabolic adaptation, and nitrogen balance in adults (aged ≥45 years) with overweight/obesity receiving weekly Incretin-Based obesity management medication treatment for 6 months.

A parallel design, open-label, multicenter randomized controlled trial will be conducted among 240 patients (aged ≥45 years) initiating Incretin-Based obesity management medication. Participants will be recruited through obesity clinics at the Tel-Aviv Sourasky Medical Center and the Tel-Aviv Assuta Medical Center, obesity clinics of HMOs, and social media groups. They will be randomly assigned to one of two groups in a 1:1 ratio: protein supplements ('Easy Whey' 25 gr protein/day) plus weekly resistance training and no intervention. Data will be collected at baseline, 3, and 6 months, including demographics, medical status, body composition, functional parameters, resting metabolic rate, nitrogen balance, and physical activity performance.

All participants will be advised to follow an exercise regime, a reduced-calorie diet based on the principle of the Mediterranean eating pattern and be encouraged to follow a regular meeting schedule with a registered dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥45 years.
* Overweight or obese (BMI ≥30, or BMI ≥27 with at least one obesity-related comorbidity).
* Eligible to receive incretin-based weight loss medications (e.g. Wegovy or Mounjaro).
* Able to read and speak Hebrew fluently.

Exclusion Criteria:

* Medical contraindications for incretin-based weight-loss medications.
* Current treatment with insulin or sulfonylurea medications.
* Inflammatory bowel disease.
* Active or unstable psychiatric disorders or cognitive impairment.
* Active bulimia nervosa.
* Previous bariatric surgery or bariatric endoscopic procedures.
* Use of other weight management medications within the past month.
* Weight loss of ≥5% within the past three months.
* Implanted cardiac pacemaker or other electronic implants.
* Regular resistance training within the past three months.
* Regular use of protein supplements.
* Allergy or intolerance to dairy proteins or vegan lifestyle.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Mass (kg) | Baseline, 3 months, 6 months.
  Change in fat mass (in kilograms) as measured by InBody 770 bioelectrical impedance analysis
Change in Fat Mass Percentage (%) | Baseline, 3 months, 6 months.
  Change in fat mass percentage (%) as measured by InBody 770 bioelectrical impedance analysis
Change in Lean Body Mass (kg) | Baseline, 3 months, 6 months.
  Change in lean body mass (in kilograms) as measured by InBody 770 bioelectrical impedance analysis.
Change in Skeletal Muscle Mass (kg) | Baseline, 3 months, 6 months.
  Change in skeletal muscle mass (in kilograms) as measured by InBody 770 bioelectrical impedance analysis.
Change in Body Mass Index (BMI) | Baseline, 3 months, 6 months.
  hange in Body Mass Index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m²), based on body weight measured by InBody 770.

SECONDARY OUTCOMES:
Change in Resting Metabolic Rate | Baseline, 3 months, 6 months.
  Changes in resting metabolic rate measured using indirect calorimetry (Q-NRG)
Change in Nitrogen Balance | Baseline, 3 months, 6 months.
  Nitrogen balance measured by 24-hour urine collection to evaluate protein usage in the body.
Change in Short Physical Performance Battery (SPPB) score | Baseline, 3 months, 6 months.
  Change in physical function assessed using the SPPB, which includes balance, gait speed, and chair stand tests.
  Unit of Measure: Score from 0 to 12; higher scores indicate better physical function.
Change in Sit-to-Stand Test Performance | Baseline, 3 months, 6 months.
  Change in the number of repetitions completed in the 30-second sit-to-stand test.
  Unit of Measure: Number of repetitions
Change in Handgrip Strength | Baseline, 3 months, 6 months.
  Change in maximal isometric handgrip strength measured using a dynamometer (e.g., JAMAR).
  Unit of Measure: Kilograms (kg)
Change in Nutrient Intake Based on 3-Day Food Diaries | Baseline, 3 months, 6 months.
  Average daily intake of protein, fat, and carbohydrates (in grams per day) derived from 3-day food diaries.
  Unit of Measure: Grams per day (g/day)
Change in Mediterranean Diet Adherence | Baseline, 3 months, 6 months.
  Assessed by the Israeli Mediterranean Diet Adherence Screener (higher scores indicate better adherence on a scale).
  Unit of Measure - Score
Change in Eating Behavior - Control of Eating Questionnaire (CoEQ) | Baseline, 3 months, 6 months.
  Change in eating behavior assessed by CoEQ; higher scores indicate greater control over eating behavior.
  Unit of Measure: Score
Change in Food Reward Sensitivity - Power of Food Scale (PFS) | Baseline, 3 months, 6 months.
  Assessed using the Power of Food Scale (higher scores reflect greater sensitivity to food cues).
  Unit of Measure: Score

IPD SHARING:
Plan to Share IPD: Undecided